CLINICAL TRIAL: NCT06658782
Title: Abbreviated Magnetic Resonance Imaging vs Ultrasound Surveillance for Liver Cancer dETection in People at High Risk of Developing Liver Cancer
Acronym: AMULET
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Bournemouth University (Other); Glasgow Caledonian University (Other); Nottingham University Hospitals NHS Trust (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 333813; 24/NW/0286 (Other: REC)
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cirrhosis; Cirrhosis Due to Hepatitis B; Cirrhosis and Chronic Liver Disease; Cirrhosis Due to Hepatitis C; Cirrhosis of the Liver; Hepatocellular Carcinoma
Keywords: SURVEILANCE; DIAGNOSTIC ACCURACY; abbreviated MRI; no contrast enhanced MRI
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- non contrast MRI AND standard of care USS: Participants undergo ultrasound every 6 months as per routine clinical care. In addition they undergo research non-contrast enhanced MRI at the same 6 monthly intervals
  Interventions: Diagnostic Test: non contrast enhanced MRI

INTERVENTIONS:
Diagnostic Test: non contrast enhanced MRI — 6 monthly non contrast enhance MRI

SUMMARY:
Aim: To use magnetic resonance imaging (MRI) scans without contrast to help improve diagnosis of liver cancer in people who are at increased risk of developing liver cancer.

Background: People with any condition that affects the liver over a long period of time can develop cirrhosis. Conditions and risk factors that can lead to cirrhosis include alcohol excess, liver steatosis (lipid or fat accumulation in the liver) and infection with the viruses hepatitis B and C. One of the concerns about people with cirrhosis is that they are at increased risk of developing liver cancer. People with cirrhosis are recommended to have an ultrasound scan (USS) every 6 months (surveillance for liver cancer) so that if a cancer develops, it is diagnosed at an early stage when it can be cured. However, ultrasound can miss cancers even in people having scans every 6 months. Furthermore, the risk of cancer is not alike among people with cirrhosis. For example, people with more advanced cirrhosis and those with cirrhosis from hepatitis B are at higher risk. It is therefore possible that better tests than ultrasound are needed for people with cirrhosis who are at particularly high risk of developing cancer.

Computed tomography (CT) and Magnetic Resonance Imaging (MRI) scans with dye injection (contrast) are used for liver cancer diagnosis. However, they cannot be done every 6 months because of costs, capacity and toxicity from high CT radiation doses, and MRI contrast build-up in the brain with repeated MRI contrast injections. MRI scans without contrast are not toxic, could be done in 20 minutes and are cheaper, so could be done every 6 months. In the experience of the study investigators, MRI without contrast may raise suspicion of liver cancer in cases missed by ultrasound, so it could be used for surveillance instead of ultrasound. This study aims to find out if it is feasible to use a quick MRI (20 minutes) without contrast as surveillance for liver cancer in people at high risk of liver cancer due to liver cirrhosis and to compare this MRI with ultrasound.

Design and Methods: The investigators will recruit 300 people at higher risk of developing liver cancer because of cirrhosis. Study participants will have an ultrasound scan every 6 months as they would in their standard clinical care and an additional 6 monthly non-contrast MRI scan for 30 months (6 visits). If the ultrasound or non-contrast MRI raises concern for a possible liver cancer, an MRI scan with contrast (with dye injection) will be done for definitive diagnosis. All participants will have an MRI with contrast at the end of 30 months (M30) to ensure that no cancers were missed. Participants will be asked to complete questionnaires to measure quality of life, anxiety, and their experience of MRI and ultrasound scans and data will be collected from their medical notes. The number of liver cancers detected by ultrasound will be compared to the number detected by the non-contrast MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study AND

  * All genders, aged 18 years or above AND
  * Eligible for HCC US surveillance in the opinion of the local investigators AND
  * Child Pugh score A or B AND
  * Diagnosed with liver cirrhosis due to ArLD, MASLD, chronic hepatitis C, chronic hepatitis B, genetic haemochromatosis AND
  * Have an annual risk of HCC of at least 3% as determined by the aMAP score OR
  * Participants with chronic liver disease (with or without cirrhosis) who had successful treatment for HCC, have not had a recurrence and have returned to 6 monthly surveillance with USS

Exclusion Criteria:

* • Contraindication to MRI

  * Known allergy / reaction to intravenous gadolinium contrast
  * Prisoners
  * Pregnancy or breast feeding
  * Previous liver transplant
  * Participants who are known to have indeterminate liver nodules on prior imaging requiring ongoing follow-up with MRI or CT
  * Previous HCC treated with curative intent and still being followed up with CT or MRI with contrast for possible recurrence
  * Estimated glomerular filtration rate of <30 ml/min/1.73m2
  * Participant is on haemodialysis
  * Participants who are unlikely to comply with the study procedures in the opinion of the local investigator
  * In the view of the clinician, if the participant has a co-morbidity likely to lead to death within the following 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a high risk of HCC will be included. Participants will have liver cirrhosis from Alcohol related liver disease, metabolic dysfunction associated steatotic liver disease, chronic hepatitis C, chronic hepatitis B or genetic haemochromatosis, or with chronic liver disease and prior successful treatment for HCC without recurrence and who are back in surveillance with USS.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2039-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance for HCC | from enrolment to 30 months
  True positive tests for HCC per round of surveillance False positive tests for HCC per round of surveillance Positive predictive value for HCC per round of surveillance True negative tests for HCC over the 30 months of surveillance False negative tests for HCC over the 30 months of surveillance Sensitivity and specificity of nceMRI and USS for HCC over 30 months of surveillance

SECONDARY OUTCOMES:
stage and size of HCC at diagnosis | from enrolment to 30 months
  Numbers of HCC detected by nceMRI and USS at a very early, early, intermediate or advanced stage as defined by the Barcelona Clinic Liver Cancer staging system.
  The number and size of HCC tumours per participant with HCC The number of new indeterminate lesions identified at each surveillance round
proportion of participants that receive treatment with curative intent | from enrolment to 30 months
  Proportion of participants diagnosed with HCC who go on to receive treatment with curative intent
Quality of Life, Anxiety and Depression | from enrolment to 30 months
  Results of the EQ-5D-5L questionnaire and Hospital Anxiety and Depression Scale questionnaire
participant experience | baseline, and month 24
  Results of participant experience questionnaire
number of unused appointments | from enrolment to 30 months
  We will count how many appointments for HCC surveillance are unused due to appointments that are missed by participants or cancelled buy the health care provider, or due to participants being lost to follow-up or participants where HCC surveillance is no longer indicated.
multivariate models | month 30
  Sensitivity and specificity of multivariable models for the diagnosis of HCC
mechanistic sub-study quantitative MRI metrics | from baseline to months 30
  Quantitative variables extracted from MRI data; T1 (ms), R2* (ms), PDFF (%), ADC (mm2/s)
long term outcomes | Up to 10 years after the last study MRI scan is performed
  A composite end point including the outcomes of: all cause mortality, liver related mortality, liver decompensation (ascites, hepatic encephalopathy, variceal bleeding), hepatocellular cancer, non primary liver cancer, liver transplantation.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trudt, Oxford, Oxon
  - Bournemouth University Hospital, Bournemouth

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be shared with global academic, commercial or other collaborators after analysis and publication of results, which is expected to be after the end of the study.